CLINICAL TRIAL: NCT03879109
Title: A Phase III Randomized Trial Evaluating Chemotherapy Followed by Pelvic Reirradiation Versus Chemotherapy Alone as Pre-operative Treatment for Locally Recurrent Rectal Cancer (GRECCAR - PRODIGE - FRENCH)
Brief Title: Chemotherapy Followed by Pelvic Reirradiation Versus Chemotherapy Alone as Pre-operative Treatment for Locally Recurrent Rectal Cancer
Acronym: GRECCAR15
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2017/52
Record Dates: First submitted 2019-03-13; First posted 2019-03-18 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Rectal Cancer
Keywords: Locally recurrent rectal cancer; Pelvic reirradiation; Oncological surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Induction Chemotherapy followed by Pelvic reirradiation (Experimental): Protocol of chemotherapy FOLFIRINOX*, 6 cycles :
  * oxaliplatin: 85 mg/m2
  * irinotecan: 180 mg/m²
  * folinic acid: 400 mg/m2
  * 5FU : 400 mg/m2 (bolus)
  * 5FU : 2400 mg/m2 (continuous infusion)
  Protocol of reirradiation consists in conformational intensity modulated external irradiation, delivering a 30.6 Gy dose (1.8 Gy/day), with concomitant chemotherapy including Capecitabine 1600 mg/m²/day, five days a week.
  Interventions: Drug: Chemotherapy FOLFIRINOX, 6 cycles; Radiation: Radiochemotherapy; Procedure: Surgery
- Arm B: Chemotherapy alone (Active Comparator): Protocol of chemotherapy FOLFIRINOX*, 6 cycles :
  * oxaliplatin: 85 mg/m2
  * irinotecan: 180 mg/m²
  * folinic acid: 400 mg/m2
  * 5FU : 400 mg/m2 (bolus)
  * 5FU : 2400 mg/m2 (continuous infusion)
  Interventions: Drug: Chemotherapy FOLFIRINOX, 6 cycles; Procedure: Surgery

INTERVENTIONS:
Drug: Chemotherapy FOLFIRINOX, 6 cycles — * oxaliplatin: 85 mg/m2
  * irinotecan: 180 mg/m²
  * folinic acid: 400 mg/m2
  * 5FU : 400 mg/m2 (bolus)
  * 5FU : 2400 mg/m2 (continuous infusion)
Radiation: Radiochemotherapy — Reirradiation consists in conformational intensity modulated external irradiation (Intensity-modulated radiotherapy Volumetric Modulated Arc Therapy or tomotherapy) delivering a 30.6 Gy dose with high-energy photons in fractions of 1.8 Gy per day (17 fractions) 5 days a week With Concomitant chemotherapy including Capecitabine 1600 mg/m²/day, five days a week.
  Arms: Arm A: Induction Chemotherapy followed by Pelvic reirradiation
Procedure: Surgery — Surgery will be performed at:
  * Arm A: 8 weeks (±1) after the end of treatment
  * Arm B: 6 weeks (±1) after the end of treatment
  Surgical procedures are defined into three categories:
  * Total mesorectal excision (TME)
  * Extended-TEM (e-TME)
  * Pelvic exenteration (PE)

SUMMARY:
GRECCAR 15 is focused on Locally Recurrent Rectal Cancer (LRRC) for patients with previous pelvic radiotherapy for the primary rectal cancer. This situation leads to a 20% higher risk of non-curative resection for the LRRC management (R1 status) impacting significantly the overall survival. The widespread use of neoadjuvant radiotherapy for primary rectal cancer introduces this new problem: the treatment of LRRC in previously irradiated area.

The objective of GRECCAR 15 is to assess the efficacy of neoadjuvant chemotherapy followed by pelvic reirradiation versus neoadjuvant chemotherapy alone on the rate of curative surgery (R0) in previously irradiated patients with LRRC.

DETAILED DESCRIPTION:
The incidence of rectal cancer in the European Union is 15-25/100 000 per year. There is a 5-10% rate of locally recurrent rectal cancer (LRRC), with an overall survival rate of 40% at 5 years after complete resection. Curative surgery of LRRC requires multi-visceral resections which are associated with significant post-operative morbidity of 60%. Despite the combination of a potential curability and the high post-operative morbidity, there are currently neither good data from prospective randomized studies regarding optimum preoperative treatments for LRRC nor is there data assessing the efﬁcacy of response to any such treatments. Moreover, the widespread use of neoadjuvant radiotherapy for primary cancer introduced a new problem: the treatment of LRRC in previously irradiated area. Some studies investigated various modalities of reirradiation and showed acceptable late toxicity and encouraging outcome. GRECCAR 15 would be the first prospective randomized trial so far to evaluate the interest of pelvic reirradiation for LRRC, in previously irradiated patients.

The objective is to assess the efficacy of neoadjuvant chemotherapy followed by pelvic reirradiation versus neoadjuvant chemotherapy alone on the rate of curative surgery (R0) in previously irradiated patients with LRRC.

Patients will be followed every 4 months during 2 years, and every 6 months the last year with chest, abdominal and pelvic scan and tumour markers.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Age ≥18 years
* LRRC (histologically proven) ≤ 15 cm from the anal verge
* First or second LRRC (histologically proven) ≤ 15 cm from the anal verge
* Previous pelvic irradiation for the primary rectal cancer or primary recurrence (25-50.4Gy)
* No distant metastasis
* Resectable locally recurrent rectal cancer (according to the International consensus, absolute contraindications for resectabililty are bilateral sciatic nerve involvement, circumferential bone involvement, high sacral involvement requiring total sacrectomy; relative contraindications for resectabilty are sciatic notch involvement and encasement external iliac vessels)
* Adequate hematologic function : Hemoglobin ≥ 9 g/dL, leukocytes ≥ 4000/mm3, neutrophil count ≥ 1500/mm3, blood platelets ≥ 100 000/mm3
* Adequate hepatic function : total bilirubin ≤ 1,5 x ULN, ASAT et ALAT ≤ 3 x ULN, alkalin phosphatases ≤ 3 x ULN
* Adequate renal function : creatinine clearance ≥ 30 ml/min
* ECOG performance status < 2
* Women not sterilized by the first treatment (ovarian transposition) and males (and their female partners) patients agree to use two methods of effective contraception (one of them being a barrier method) during the study, for at least 6 months for men and for women after the last administration of study treatment
* Patient affiliated to a social security system or beneficiary of the same
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Recurrent rectal cancer after local excision
* Concomitant cancer or medical history of cancer within 5 years other than cancers treated in situ (cervical carcinoma or basocellular carcinoma or spinocellular carcinoma)
* Contraindication for chemotherapy Contraindication for chemotherapy (refer to Summary of characteristics of the products of the study drugs available at http://base-donnees-publique.medicaments.gouv.fr) or radiotherapy or surgery
* Symptomatic cardiac or coronary insufficiency
* Personal or family history of long QT syndrome congenital
* ECG at screening or baseline (predose) with QT/QTc > 450 msec (male) or QT/QTc > 470 msec (female)
* Chronic inflammatory bowel disease and/or bowel obstruction
* Patients with hypocalcemia, hypokalemia, hypomagnesemia.
* Progressive active infection (HIV or chronic hepatitis B or C) or any other severe medical condition that may preclude the delivery of treatment
* Complete or partial Dihydropyrimidine deshydrogenase (DPD) deficiency (uracilemia ≥ 16 ng/mL)
* If contraindication to FOLFIRINOX, possibility to administred FOLFOX or FOLFIRI +/-EGFR (Contraindication to oxaliplatin: peripheral neuropathy > grade 1 (CTCAE grading system v5.0)
* Peripheral neuropathy > grade 1 (CTCAE grading system v5.0)
* Concomitant treatment with millepertuis, yellow fever vaccine, live attenuated vaccine, phenytoin, warfarin or sorivudine (or chemically equivalent)
* Pregnant or breast-feeding woman
* Persons deprived of liberty or under guardianship or incapable of giving consent
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule, as assessed by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of curative surgery | At surgery, expected average 6 to 8 weeks after neoadjuvant treatment
  To determine the rate of R0 resection

SECONDARY OUTCOMES:
Disease Free Survival | From surgery until 3 years of follow-up
  Rate of disease-free survival at 3 years
Overall Survival | From surgery until 3 years of follow-up
  Rate of overall survival at 3 years
Surgical morbidity | From surgery until 30 days after surgery
  To analyse surgical morbidity (Dindo classification) during first 30 days after the surgery
Surgical mortality | From surgery until 30 days after surgery
  To analyse surgical mortality (Dindo classification) during first 30 days after the surgery
Compliance to treatment | From beginning of neoadjuvant treatment until surgery, expected average 20 weeks after neoadjuvant treatment
  Proportion of patients receiving full allocated neoadjuvant treatment
Proportion of good tumor response | At 6 weeks (Arm A) and 4 weeks (Arm B) after neoadjuvant treatment
  Rate of tumor with a decreasing size of 50% at least after preoperative treatment at MRI
Quality of life (QLQ CR-30) | Before neoadjuvant treatment, before surgery, 4 months, one year and two years after surgery
  The scores of questionnaire QLQ C-30 will be examined The EORTC QLQ-C30 is a patients self-rating questionnaire that measures physical, role, social, emotional, and cognitive functions as well as overall QoL. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Quality of life (QLQ CR-29) | Before neoadjuvant treatment, before surgery, 4 months, one year and two years after surgery
  The scores of questionnaire QLQ CR-29 will be examined. The EORTC QLQ-CR29 has five functional and 18 symptom scales. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Tolerance to treatment | From beginning of neoadjuvant treatment until 1 year after surgery
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LAURENT, Principal Investigator — University Hospital, Bordeaux
Locations (13):
- France (13):
  - Institut Sainte Catherine, Avignon
  - CHU Bordeaux, Bordeaux
  - CHU Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Hospices Civils de Lyon, HCL, Lyon
  - Institut Paoli Calmette, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denost Q, Frison E, Salut C, Sitta R, Rullier A, Harji D, Maillou-Martinaud H, Rullier E, Smith D, Vendrely V; on behalf the GRECCAR Group. A phase III randomized trial evaluating chemotherapy followed by pelvic reirradiation versus chemotherapy alone as preoperative treatment for locally recurrent rectal cancer - GRECCAR 15 trial protocol. Colorectal Dis. 2021 Jul;23(7):1909-1918. doi: 10.1111/codi.15670. Epub 2021 Jun 10. PMID 33843133